CLINICAL TRIAL: NCT03520218
Title: A Pilot Study to Evaluate Low-Dose Positron Emission Mammography Imaging in Visualization and Characterization of Suspicious Breast Abnormalities
Brief Title: Evaluating Positron Emission Mammography Imaging of Suspicious Breast Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-5029
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Performance of R-PEM (Experimental): 5mCi of F-18 FDG will be injected and patients will wait for uptake of FDG before proceeding with first set of R-PEM scans. Additional optional R-PEM scans may be performed 4 hours after injection, and then possibly 7 hours after injection.
  These R-PEM images will be compared to standard diagnostic breast work-up using DBT and MRI
  Interventions: Device: Performance of R-PEM

INTERVENTIONS:
Device: Performance of R-PEM — R-PEM imaging will produce high-sensitivity images with low levels of F-18 FDG and optional subsequent scans performed will display reduced levels of the injected radiotracer.

SUMMARY:
The goal of this pilot project is to test the new Radialis Positron Emission Mammography (R-PEM) system in breast cancer patients that has a higher sensitivity with lower radiation doses than conventional PET/CT.

The plan for the pilot study is to image patients who are already scheduled for diagnostic imaging for breast cancer after a positive core biopsy. Participants will be injected with 5mCi (millicurie) of F18-Fluorodeoxyglucose (FDG) and patient will wait for a couple of hours for uptake of FDG. After this time, the first R-PEM scan will occur. Additional optional R-PEM scans can be performed 4 hours after injection and 7 hours after injection with reductions in radiation emission.

Additionally, R-PEM images will be compared to standard-of-care breast Magnetic Resonance Imaging (MRI) and digital breast tomosynthesis (DBT) to study extension of disease and screening of contralateral breast.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of any race and ethnicity
* Subject is at least 26 years old
* Following routine mammography imaging, subject is categorized as BI-RADS score 4C or 5 because of calcifications, masses, asymmetries or/and architectural distortion will undergo additional tests including biopsy within 30 days of routine imaging
* Subject is female with a recent breast biopsy confirming breast cancer

Exclusion Criteria:

* Subject unable or unwilling to undergo informed consent
* Subjects who are unable or unwilling to tolerate any of the imaging tests because of claustrophobia, compression, etc.
* Subjects who are pregnant or who think they may be pregnant
* Subjects who are breast-feeding
* Subjects weight exceed table limits of MRI and PET-CT (300-450 lb or 135-205 kg)
* Subjects with history of allergic reaction to gadolinium or previous history of life-threatening anaphylactic reaction to any contrast.
* Claustrophobic subjects

Min Age: 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Evaluating Performance of the R-PEM system as the Dose Decays | 2 years
  The diagnostic performance of R-PEM including sensitivity, specificity, positive and negative predictive values compared to magnetic resonance imaging, digital breast tomosynthesis mammography, and digital mammography in characterization of suspicious breast abnormalities will also be evaluated in our study when those images are available through standard patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Vivianne Freitas, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, University Health Network, 610 University Ave., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Freitas V, Li X, Scaranelo A, Au F, Kulkarni S, Ghai S, Taeb S, Bubon O, Baldassi B, Komarov B, Parker S, Macsemchuk CA, Waterston M, Olsen KO, Reznik A. Breast Cancer Detection Using a Low-Dose Positron Emission Digital Mammography System. Radiol Imaging Cancer. 2024 Mar;6(2):e230020. doi: 10.1148/rycan.230020. PMID 38334470